CLINICAL TRIAL: NCT00655577
Title: Role of Exercise in Prevention of Osteoporotic Fractures in Elderly Women
Brief Title: Exercise and Prevention of Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Ministry of Education (Ambiguous); Juho Vainio Foundation (Other); Miina Sillanpää Foundation (Unknown); Finnish Cultural Foundation (Other); Oulu Deaconess Institute (Other); Northern Ostrobothnia District Hospital (Unknown)
Responsible Party: Raija Korpelainen, Oulu Deaconess Institute, Department of Sports Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K78751
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Bone Mineral Density; Strength; Balance; Osteoporosis; Fractures
Keywords: Aging; Osteoporosis; Exercise; Population based; Randomized trial; Falls; Fractures
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Control group
  Interventions: Behavioral: Exercise
- 1 (Experimental): Exercise group
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Supervised, mainly home-based balance, strength and jumping exercises

SUMMARY:
The significance of this population-based study is in producing new information for planning interventions and rehabilitation programs for the elderly, planning education of health care personnel and planning national health education programs for different age groups.

The study consists of an epidemiological cross-sectional study and a randomized controlled intervention study. The study population consisted of all the 1689 home-dwelling women born during 1924-1927 residing in Oulu, Northern Finland, who were asked to a screening visit including bone mineral density (BMD) measurement of the distal radius in 1997. 1222 women attended the clinic and were afterwards mailed a postal questionnaire focusing on lifelong risk factors for osteoporosis, e.g. the amount of physical activity at work and during leisure time, daily intake of calcium and use of alcohol and cigarettes. Those with BMD value more than 20% lower than the reference value, underwent a densitometry of the hip. All women with femoral neck BMD more than 20% below the reference value (n=160) were randomly selected to either exercise (n=84) or control (n=76) group. At baseline and after that annually during the 30-month intervention, balance, muscle strength, aerobic capacity, walking speed, cognitive functions and mood are measured from all the participants. Hip BMD will be measured annually. The exercise group participates in a supervised training program with weekly sessions from the beginning of October to the end of April. In addition to the supervised sessions the participants train daily at home. From April to October the exercises are performed purely at home. The training regimen consists of balance, strength and impact exercises. The intervention group keeps diary of their daily physical activity. The number and severity of falls are recorded from both the groups.

The purpose of the study is:

1. to identify factors accounting for low BMD in elderly home-dwelling women with severe osteopenia.
2. to evaluate how supervised regular weight-bearing exercise program affects BMD in elderly home-dwelling women with severe osteopenia
3. to evaluate how supervised regular balance and muscle training affects balance and muscle strength in elderly home-dwelling women with severe osteopenia.

   In addition the aim is to:
4. study how regular supervised exercise affects the incidence and severity of falls, mood and cognitive functions in women with severe osteopenia.

Hypothesis and research methods

The main hypothesis is that long-term supervised, mainly home- based regular impact-type and balance and muscle exercises can improve balance and muscle strength of lower extremities and maintain bone mass in elderly women. We also hypothesize that the incidence of falls is lower in the exercise group than in the controls and that the falls are more injurious in the control group than in the intervention group during the follow-up period

ELIGIBILITY:
Inclusion Criteria:

* female gender
* born during 1924-1927 and living in Oulu, Finland in 1997
* distal radius BMD value of more than 2 SD below the reference value
* hip BMD value of more than 2SD below the reference value

Exclusion Criteria:

* use of walking aid device other than a stick
* bilateral hip joint replacement
* unstable chronic illness
* malignancy
* medication known to affect bone density
* severe cognitive impairment
* involvement in other interventions

Ages: 71 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 1998-08; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sirkka Keinänen-Kiukaanniemi, MD,PhD, Study Director — University of Oulu, Department of Public Health Sciences and General Practice
Locations (1):
- Oulu Deaconess Institute, Department of Sports Medicine, Oulu, Finland

REFERENCES:
- [Derived] Korpelainen R, Keinanen-Kiukaanniemi S, Nieminen P, Heikkinen J, Vaananen K, Korpelainen J. Long-term outcomes of exercise: follow-up of a randomized trial in older women with osteopenia. Arch Intern Med. 2010 Sep 27;170(17):1548-56. doi: 10.1001/archinternmed.2010.311. PMID 20876406